CLINICAL TRIAL: NCT06284694
Title: Treatment of Neuropathic Pain Following Spinal Cord Injury - a Repetitive Transcranial Magnetic Stimulation Approach
Brief Title: Treatment of Neuropathic Pain Following Spinal Cord Injury - a RTMS Approach
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB23-0120
Record Dates: First submitted 2024-02-14; First posted 2024-02-29 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-02

CONDITIONS: Neuropathic Pain
Keywords: Spinal Cord Injury
MeSH Terms: conditions — Neuralgia; Spinal Cord Injuries | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: All participants will receive active rTMS treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Repetitive Transcranial Magnetic Stimulation (rTMS) (Experimental): Participants will undergo high frequency rTMS sessions 5 days a week for 4 weeks (20 treatments total). Treatment intensity will be applied at 100-120% of the participant's resting motor threshold. The neurostimulation protocol will be 10 trains of 60 pulses (600 pulses total) at a frequency of 10 Hz, with inter-train interval of 45-seconds. The rTMS will be administered to the dorsolateral prefrontal cortex (DLPFC) which will be located using Montreal Neurologic Institute (MNI) coordinates (-50, 30, 36) on a standardized brain. Participants will be seated in a comfortable chair or their wheelchair for each rTMS session.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — See experimental arm description

SUMMARY:
This study aims to determine if repetitive transcranial magnetic stimulation (rTMS) can improve pain symptomology in adults with neuropathic pain (NP) following a spinal cord injury (SCI).

DETAILED DESCRIPTION:
Approximately 86,000 Canadians live with a spinal cord injury (SCI). Individuals with a SCI experience varying levels of deficits in motor and sensory function and sometimes paralysis. SCI can result in permanent impairments both physical and psychological, as the loss of body function greatly impacts quality of life. Neuropathic pain (NP) is a common complication following SCI. Damage or dysfunction to the nervous system after SCI commonly leads to secondary injury or disease in the somatosensory system, which may contribute to NP. This debilitating complication can impede many factors including physical function, rehabilitation, sleep, and return to work.

Treatment modalities for NP aim to reduce pain and improve function and quality of life. Pharmacological interventions are considered first-line therapy for NP management, though there remains limited evidence to support the efficacy of this treatment modality. Pharmacologic therapies may also include negative side effects. Additionally, clinical guidelines for NP management recommend including non-pharmacologic strategies. Therefore, an interdisciplinary strategy may be required to effectively mitigate NP after SCI. Evidence of neuromodulation techniques to improve various pain conditions is well established, and reductions in pain may be related to the modified brain activity. Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive neuromodulation intervention with a low risk of adverse effects. Preliminary studies investigating rTMS for NP after SCI have shown a therapeutic effect after treatment whereby quality of life and pain improved in this population.

RESEARCH QUESTION AND OBJECTIVES

This study aims to determine the clinical feasibility of a rTMS protocol to improve pain symptomology in adults with NP following SCI. Additionally, this study will contribute to the limited body of evidence for the efficacy of this treatment modality in this population.

The primary objective is to determine symptomatic changes in pain profile and treatment response using the International Spinal Cord Injury Pain Basic Data Set (ISCIPBDS) self-report version, a valid and reliably tested instrument, and the PROMIS Scale Neuropathic Pain Quality 5a questionnaire.

Secondary objectives include assessing quality of life (QLI-SCI), depression (PHQ-9), anxiety (GAD-7), disability (WHODAS), and pain catastrophizing (PCS).

METHODS

Clinical Assessments: Demographic information, including age, sex, gender, and past medical history will be collected prior to participation. Participant's neurological level of impairment will be determined by a treating physician, allied health professional, or research study physician. The initial assessment will include answering questionnaires: International Spinal Cord Injury Pain Basic Data Set (ISCIPBDS) self-report version, PROMIS Scale Neuropathic Pain Quality 5a questionnaire, Quality of Life Index Spinal Cord Injury v3 (QLI-SCI), Pain Catastrophizing Scale (PCS), World Health Organization Disability Assessment Schedule (WHODAS) 2.0, Generalized Anxiety Disorder scale-7 (GAD-7), Patient Health Questionnaire-9 (PHQ-9), and previous medication and treatment questionnaires. Participant's current medication usage will be monitored during the study and rTMS tolerability will be assessed immediately following each treatment session. Participants will be asked to complete the above-mentioned questionnaires post-rTMS treatment, at 1 and 3 months after their last rTMS treatment.

TMS Protocol: Participants will undergo high frequency rTMS sessions 5 days a week for 4 weeks (20 treatments total). Daily rTMS sessions will include 10 trains of 60 pulses (600 pulses total) at a frequency of 10 Hz, with an inter-train interval of 45-seconds. Treatment intensity will be applied at 100-120% of the participant's resting motor threshold (RMT). A RMT is the minimal intensity required to evoke a motor evoked potential and will be obtained by administering single-pulse TMS to the left motor cortex. Electromyography (EMG) electrodes will be placed on the contralateral abductor pollicis brevis (APB) muscle to determine the motor evoked potential peak-to-peak amplitude, requiring 50 microvolts amplitude in 5 of 10 consecutive stimulations. The rTMS treatment will be administered to the dorsolateral prefrontal cortex (DLPFC) which will be located using Montreal Neurologic Institute (MNI) coordinates (-50, 30, 36). Participants will be seated in a comfortable chair or their wheelchair for each rTMS session.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed spinal cord injury
* Neuropathic pain for at least 3-months, as diagnosed by a physician
* Pain not attributable to any other conditions
* Aged 18-75 years
* Can complete wheelchair transfers independently

Exclusion Criteria:

* Prior history of transcranial magnetic stimulation (TMS) therapy
* Any TMS-related contraindications, for example: pacemaker, metallic implant, other medical conditions such as structural brain disease, previous seizure, psychiatric disorders (excluding depression and anxiety), suicide attempt in the past 6 months, liver or kidney disease, malignancy, uncontrolled hypertension or diabetes, and current pregnancy or the desire to become pregnant in the next 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
International Spinal Cord Injury Pain Basic Data Set (ISCIPBDS) self-report version | To be assessed at baseline, after rTMS treatment (1-month), and at 1-month and 3-months after rTMS treatment.
  Pain profile, including location, intensity, and interference over the past 7 days will be assessed using the ISCIPBDS self-report tool.
Patient-Reported Outcomes Measurement Information System (PROMIS) Scale Neuropathic Pain Quality 5a | To be assessed at baseline, after rTMS treatment (1-month), and at 1-month and 3-months after rTMS treatment.
  Neuropathic pain will be assessed using the PROMIS Scale Neuropathic Pain Quality 5a questionnaire. This tool assesses 5 descriptors of neuropathic pain quality. Participants are asked to rate their pain quality from 1(not at all) to 5 (very much) using a recall period of the past 7 days.

SECONDARY OUTCOMES:
Quality of Life Index Spinal Cord Injury version (QLI-SCI) | To be assessed at baseline, after rTMS treatment (1-month), and at 1-month and 3-months after rTMS treatment.
  Quality of life and satisfaction with aspects of quality of life will be assessed using the QLI-SCI instrument. This questionnaire focuses on the categories of health and functioning, social and economic, psychological/spiritual, and family.
Pain Catastrophizing Scale (PCS) | To be assessed at baseline, after rTMS treatment (1-month), and at 1-month and 3-months after rTMS treatment.
  Pain experience will be assessed using the PCS. Participants are asked to rate how much they agree with the listed thoughts and feelings they may have when experiencing pain from 0 (not at all) to 4 (all the time).
World Health Organization Disability Assessment Schedule (WHODAS) 2.0 | To be assessed at baseline, after rTMS treatment (1-month), and at 1-month and 3-months after rTMS treatment.
  Health and disability will be assessed using the WHODAS 2.0 instrument. Participants will be asked to rate the amount of difficulty that have had completing activities over the past 30 days using the scale none to extreme or cannot do.
Generalized Anxiety Disorder scale-7 (GAD-7) | To be assessed at baseline, after rTMS treatment (1-month), and at 1-month and 3-months after rTMS treatment.
  Anxiety will be assessed using the GAD-7 tool. Participants will rate the frequency of anxious feelings from 0 (not at all) to 3 (nearly every day), thinking back over the past 2 weeks. Higher scores will indicate a greater severity of anxiety symptoms.
Patient Health Questionnaire-9 (PHQ-9) | To be assessed at baseline, after rTMS treatment (1-month), and at 1-month and 3-months after rTMS treatment.
  Depression will be assessed using the PHQ-9 tool. Participants will rate the frequency of depressive thoughts and/or feelings experienced over the past 2 weeks from 0 (not at all) to 3 (nearly every day). Higher scores will indicate a greater severity of depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Chantel T Debert, MD MSc FRCPC, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burke D, Fullen BM, Stokes D, Lennon O. Neuropathic pain prevalence following spinal cord injury: A systematic review and meta-analysis. Eur J Pain. 2017 Jan;21(1):29-44. doi: 10.1002/ejp.905. Epub 2016 Jun 24. PMID 27341614
- [Background] Hatch MN, Cushing TR, Carlson GD, Chang EY. Neuropathic pain and SCI: Identification and treatment strategies in the 21st century. J Neurol Sci. 2018 Jan 15;384:75-83. doi: 10.1016/j.jns.2017.11.018. Epub 2017 Nov 16. PMID 29249383
- [Background] Almeida C, Monteiro-Soares M, Fernandes A. Should Non-Pharmacological and Non-Surgical Interventions be Used to Manage Neuropathic Pain in Adults With Spinal Cord Injury? - A Systematic Review. J Pain. 2022 Sep;23(9):1510-1529. doi: 10.1016/j.jpain.2022.03.239. Epub 2022 Apr 10. PMID 35417793
- [Background] Shen Z, Li Z, Ke J, He C, Liu Z, Zhang D, Zhang Z, Li A, Yang S, Li X, Li R, Zhao K, Ruan Q, Du H, Guo L, Yin F. Effect of non-invasive brain stimulation on neuropathic pain following spinal cord injury: A systematic review and meta-analysis. Medicine (Baltimore). 2020 Aug 21;99(34):e21507. doi: 10.1097/MD.0000000000021507. PMID 32846761
- [Background] Saleh C, Ilia TS, Jaszczuk P, Hund-Georgiadis M, Walter A. Is transcranial magnetic stimulation as treatment for neuropathic pain in patients with spinal cord injury efficient? A systematic review. Neurol Sci. 2022 May;43(5):3007-3018. doi: 10.1007/s10072-022-05978-0. Epub 2022 Mar 3. PMID 35239053
- [Background] Treede RD, Jensen TS, Campbell JN, Cruccu G, Dostrovsky JO, Griffin JW, Hansson P, Hughes R, Nurmikko T, Serra J. Neuropathic pain: redefinition and a grading system for clinical and research purposes. Neurology. 2008 Apr 29;70(18):1630-5. doi: 10.1212/01.wnl.0000282763.29778.59. Epub 2007 Nov 14. PMID 18003941
- [Background] Sun X, Long H, Zhao C, Duan Q, Zhu H, Chen C, Sun W, Ju F, Sun X, Zhao Y, Xue B, Tian F, Mou X, Yuan H. Analgesia-enhancing effects of repetitive transcranial magnetic stimulation on neuropathic pain after spinal cord injury:An fNIRS study. Restor Neurol Neurosci. 2019;37(5):497-507. doi: 10.3233/RNN-190934. PMID 31381538
- [Background] Seminowicz DA, Moayedi M. The Dorsolateral Prefrontal Cortex in Acute and Chronic Pain. J Pain. 2017 Sep;18(9):1027-1035. doi: 10.1016/j.jpain.2017.03.008. Epub 2017 Apr 8. PMID 28400293
- [Background] Brighina F, Piazza A, Vitello G, Aloisio A, Palermo A, Daniele O, Fierro B. rTMS of the prefrontal cortex in the treatment of chronic migraine: a pilot study. J Neurol Sci. 2004 Dec 15;227(1):67-71. doi: 10.1016/j.jns.2004.08.008. PMID 15546593